CLINICAL TRIAL: NCT02055846
Title: Analysis of the Mechanisms of Actions of Hsp27 Responsible of the Androgen-independent Evolution in Prostate Cancer
Brief Title: Analysis of the Mechanisms of Actions of Heat Shock Protein (Hsp27) Responsible of the Androgen-independent Evolution in Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient biological material for analysis
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PPPR / IPC 2012-002
Record Dates: First submitted 2012-10-26; First posted 2014-02-05 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2012-12

CONDITIONS: Androgen-independent Prostate Cancer
Keywords: Androgen-independent prostate cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prostate cancer (Experimental): Realisation of blood sample, urinary sample and tumor biopsy
  Interventions: Procedure: Realisation of blood sample, urinary sample and tumor biopsy

INTERVENTIONS:
Procedure: Realisation of blood sample, urinary sample and tumor biopsy

SUMMARY:
Prostate cancer (PC) represents one of the most common cancers in industrialized countries. Patients with localized disease may be treated with surgery or radiation, while androgen ablation is used as first-line therapy in patients with metastatic disease. While most patients initially respond well to this hormonal therapy, they most ultimately become unresponsive and recur within 2 years as androgen-independent prostate cancer (AIPC). Recently, docetaxel-based regimens have demonstrated improved survival in men with AIPC in two different, large, phase III studies. However, the median overall survival was prolonged for only 2 or 3 months. Androgen independent (AI) progression involves variable combinations of clonal selection, adaptive up-regulation of anti-apoptotic genes, ligand-independent androgen receptor (AR) activation, alternative growth factor pathways, and immune system escape. Additional therapeutic strategies targeting molecular mechanisms mediating resistance, combined with immunotherapy must be developed. One strategy to improve therapies in advanced PC involves targeting genes that are activated by androgen withdrawal, either to delay or prevent the emergence of the resistant AI phenotype. Recently, a scientist,identified Heat Shock Protein (Hsp27) as a highly over-expressed gene in AIPC. Hsp27 knockdown using antisens oligonucleotides (ASO) and small interfering RNA (siRNA) increased apoptotic rates and enhanced hormone- and chemo-therapy in PC. She developed and patented a 2nd generation ASO targeting Hsp27 that has been licensed (investigational drug called OGX-427) and clinical trials phase I/II is currently in process in PC. Despite OGX-427 efficiency, the functional role of stress induced Hsp27 in castration or chemotherapy-induced apoptosis remains undefined. The purpose of this study is to elucidate the pathways leading to Hsp27 action in androgen-independent prostate cancer in order to 1/ Increase the pharmacological safety of OGX-427 and 2/find new specific therapeutic targets and treatment strategy for androgen-independent prostate cancer .

ELIGIBILITY:
Inclusion Criteria:

* Prostate adenocarcinoma
* Patient > 18 years old
* Patient affiliated to a social security system or benefiting from such a system
* Signed consent to participate

Exclusion Criteria:

* Patient in emergency situation, major person being the object of a legal protective measure or unable to express its consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Level of Hsp27 protein | within 24 hours
  Mechanisms of action of Hsp27 protein to elucidate the pathways leading to Hsp27 action in androgen-independent prostate cancer (AIPC) by double hybrid Sos Recruitment System (SRS)

SECONDARY OUTCOMES:
Targets for OGX-427 | within 24 hours
  Description of new specific therapeutic targets for androgen-independent prostate cancer and pharmacological safety of OGX-427

CONTACTS AND LOCATIONS:
Overall Officials: Gwénaëlle GRAVIS, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Gwénaëlle GRAVIS, MD, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr